CLINICAL TRIAL: NCT00692055
Title: Study Evaluating the Bioavailability of Naproxen 375 mg in Two Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, POZEN
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PN400-105
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PN400
  Interventions: Drug: PN400
- 2 (Active Comparator): naproxen 375 mg
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PN400 — naproxen 375 mg / esomeprazole 20 mg
  Arms: 1
Drug: Naproxen — naproxen 375 mg
  Arms: 2

SUMMARY:
We will evaluate the bioavailability of naproxen 375 mg in two formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects between 18-55 years as well as other standard inclusion criteria for a study of this nature

Exclusion Criteria:

* Standard exclusion criteria for a study of this nature

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To assess and compare the pharmacokinetics bioavailability of a single oral dose of naproxen administered in two formulations | 72-hour PK

SECONDARY OUTCOMES:
To evaluate the safety of the two treatments | entire study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States